CLINICAL TRIAL: NCT05735132
Title: A Randomized Controlled Trial Comparing the Effects of Conventional, Bar-shaped, and V-shaped Local Infiltration Anesthesia on Pain Relief and Cannulation Success Rate in Patients Requiring Radial Artery Cannulation.
Brief Title: Novel Local Infiltration Anesthesia for Radial Artery Cannulation.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, Yi Zhang, Principal Investigator, First People's Hospital of Chenzhou
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2018012
Record Dates: First submitted 2022-12-02; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Efficiency and Safey of Radial Artery Cannulation
Keywords: Radial Artery; Local Anesthesia; Cannulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Line arm (Active Comparator): Conventional line blocking is used in radial artery cannulation for local infiltration.
  Interventions: Procedure: Conventional Line-blocking
- Bar arm (Experimental): Bar-blocking is used in radial artery cannulation for local infiltration.
  Interventions: Procedure: Bar-blocking
- V arm (Experimental): V-blocking is used in radial artery cannulation for local infiltration.
  Interventions: Procedure: V-blocking

INTERVENTIONS:
Procedure: Conventional Line-blocking — Participants will receive a 2 cm subcutaneous 1% lidocaine local infiltration injection parallel to the arm at the puncture site.
  Other Names: lidocaine infiltration at the point
  Arms: Line arm
Procedure: Bar-blocking — Participants will receive a bar-shaped subcutaneous 1% lidocaine local infiltration injection in the vertical arm, 2 cm away from the puncture site.
  Other Names: lidocaine infiltration with a cross bar
  Arms: Bar arm
Procedure: V-blocking — Participants will receive a V-shaped subcutaneous 1% lidocaine local infiltration injection at a 90-degree angle 2 cm away from the puncture site.
  Other Names: lidocaine infiltration with v shape
  Arms: V arm

SUMMARY:
This clinical trial aims to compare the pain scores and cannulation success rates of conventional, bar-shaped, and V-shaped local infiltration anesthesia in participants' radial artery cannulation.

The main questions it aims to answer are:

* Are bar-shaped and V-shaped more successful than the conventional block in radial artery cannulation?
* Are bar-shaped and V-shaped less painful than the conventional block in radial artery cannulation? Participants will describe their pain score during their radial artery cannulation.

Researchers will compare the pain scores and cannulation success rates in bar-shaped, V-shaped, and conventional line blocking to see if bar-shaped and V-shaped blocking is better choices than conventional line blocking.

DETAILED DESCRIPTION:
The purpose of the study, as well as the necessity, benefits, and risks of arterial cannulation, and the purpose of the study, were explained in detail to all participants screened by inclusion and exclusion criteria, and signed informed consent was obtained on the day before the operation.

Upon entering the operating room, participants will be connected to a pulse oximeter, noninvasive blood pressure monitor, and electrocardiograph and will record baseline heart rate, blood pressure, depth of the radial artery at the first wrist stripe before local anesthesia, and PVDF capacitance difference.

The arterial pressure transducer and tubing will be flushed with 25 U/mL of heparin saline and kept in a ready state.

Anesthesiologists not participating in the study will then be asked to open an opaque sealed envelope to determine the type of local anesthesia to be used during intubation. The conventional approach is to complete a 2 cm subcutaneous injection with 2% lidocaine directly above the artery in the direction of the palpable beat; the bar-blocking is to complete a 2 cm subcutaneous injection perpendicular to the arterial beat line 2 cm from the proximal segment of the puncture site, and the V-blocking is to complete a subcutaneous injection at a 90-degree angle with a 2-cm margin toward the distal end at 2 cm proximal to the puncture site. Heart rate, blood pressure, depth of the radial artery at the first wrist stripe, and PVDF capacitance difference were recorded at the end of local anesthesia.

The radial artery cannula will be placed with a 20 gauge radial artery catheter by palpation under the supervision of an anesthesia consultant in the operating room by another anesthesiology resident not involved in the study.

The participator's arm will be slightly abducted (less than 90 degrees) and placed on the arm board, placing the wrist in the extended position by placing a padded towel under the wrist. The wrist will then be secured to the arm board with tape. To maintain sterility, the wrist will be pretreated with 10% povidone-iodine, and surgical gloves and a sterile cloth will be used. The timer will start counting when the operator starts palpating the radial artery pulse. Immediately after successful cannulation, the assistant will connect a pressure monitoring tube. The timer will stop as soon as the arterial waveform appears on the monitor. The number of cannulations is also recorded, with one cannulation recorded for each skin puncture or each change of the puncture needle direction. If cannulation fails three times or if the radial artery is not cannulated after 360 seconds, the procedure will be aborted and recorded as "failed cannulation". A senior anesthesiologist will then complete the arterial cannulation using whatever method he/she decides. The time taken for cannulation is recorded, as well as the application of ultrasonography to measure the depth of the puncture site at the first wrist stripe after local anesthesia and the difference in PVDF membrane capacitance.

Systolic and diastolic blood pressures and heart rates were collected at the start and end of cannulation in the other arm, the time to successful placement of the radial artery cannula (in seconds), and the times of cannulation.

ELIGIBILITY:
Inclusion Criteria:

* The participant is scheduled for elective surgery.
* The participant's elective surgery required radial artery cannulation.
* Participants should be at least 18 years old.

Exclusion Criteria:

* The Allen test of the participant is negative.
* The participant has a history of peripheral vascular disease.
* The participant has a cannula site infection or lesion.
* The participant is on vasoactive medication.
* A history of artery cannulation at the planned cannulation site within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS score | upto 10 minutes
  The visual analogue scale (VAS) will evaluate pain intensity during radial artery cannulation. This scale is a 10-cm horizontal line with terminal descriptors of 0 (no pain) and 10 (worst imaginable pain) .
Time spent on radial artery cannulation | upto 5 minutes
  From the completion of local infiltration anesthesia to the completion of radial artery cannulation, up to 15 minutes.
Success rate of radial artery cannulation | upto 3 months
  Success rate will be recorded to evaluate the influences of local anesthesia to radial artery cannulation.

SECONDARY OUTCOMES:
Depth of tested radial artery | upto 5 minutes
  Depth of tested radial artery will be recorded to evaluate the influences of local anesthesia to radial artery cannulation.
Polyvinylidene fluoride (PVDF) capacitance difference | upto 5 minutes
  PVDF capacitance difference will be recorded to evaluate the influences of local anesthesia to radial artery cannulation.
Heart rate | upto 5 minutes
  Heart rate changes will be recorded to supplementally evaluate the pain intensity during the cannulation.
Blood Pressure | upto 5 minutes
  Blood Pressure changes will be recorded to supplementally evaluate the pain intensity during the cannulation.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zeng, Master, Study Chair — First People's Hospital of Chenzhou
Locations (1):
- Chenzhou First People's Hospital, Chenzhou, Hunan, China

IPD SHARING:
Plan to Share IPD: No